CLINICAL TRIAL: NCT01237444
Title: A Phase 3, Randomized, Open Label, Controlled Study of Lopinavir/Ritonavir and Lamivudine Versus Standard Therapy in Naïve HIV-1 Infected Subjects.
Brief Title: Study of Lopinavir/ Ritonavir and Lamivudine Versus Standard Therapy in Naïve HIV-1 Infected Subjects.
Acronym: GARDEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pedro Cahn (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Pedro Cahn, MD, Fundación Huésped
Organization: Fundación Huésped (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FH-10 GARDEL study
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infection
Keywords: Lopinavir/ritonavir plus 3TC as a dual therapy regimen.
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lopinavir/ritonavir plus lamivudine (Experimental): ARM 1:
  Lopinavir/ritonavir 200mg/50mg 2 tabs bid plus 3TC 150mg x1 tab bid
  Interventions: Drug: lopinavir/ritonavir plus one nucleoside
- lopinavir/ritonavir plus two nucleosides (Active Comparator): ARM 2:
  3TC 150mg x1 tab bid or FTC 200mg 1 capsule qd plus Lopinavir/ritonavir 200mg/50mg 2 tabs BID plus a second NRTI, selected at investigator's discretion, based on baseline genotype
  Interventions: Drug: lopinavir /ritonavir plus two nucleosides

INTERVENTIONS:
Drug: lopinavir/ritonavir plus one nucleoside — ARM 1:
  Lopinavir/ritonavir 200mg/50mg 2 tabs bid plus 3TC 150mg x1 tab bid
  Arms: lopinavir/ritonavir plus lamivudine
Drug: lopinavir /ritonavir plus two nucleosides — ARM 2:
  3TC 150mg x1 tab bid or FTC 200mg 1 capsule qd plus Lopinavir/ritonavir 200mg/50mg 2 tabs BID plus a second NRTI, selected at investigator's discretion, based on baseline genotype.
  Arms: lopinavir/ritonavir plus two nucleosides

SUMMARY:
The purpose of this study is designed to compare the safety, tolerability, antiviral activity and immunological effect of lopinavir/ritonavir plus lamivudine (3TC) versus standard therapy with 2 nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) plus lopinavir/ritonavir in the treatment of naïve HIV-1 infected subjects.

DETAILED DESCRIPTION:
Combination therapy with 2 nucleoside reverse transcriptase inhibitors (NRTI) plus a non-nucleoside reverse transcriptase inhibitor (NNRTI) or a protease inhibitor (PI) has been the mainstay of therapy for over 10 years, based on sound evidence derived from randomized controlled clinical trials and epidemiological data.A variety of new approaches designed to address the problems associated with combination highly active antiretroviral therapy (HAART) are currently being explored. These include strategic treatment interruptions to reduce time on therapy, toxicity and cost;Based on its performance, a dual drug combination that includes lopinavir/ritonavir and spares the more toxic NRTIs such as thymidine nucleoside-analogs, but maintains non-thymidine nucleoside-analogs appears as a potentially simple, safe and effective regimen.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age.
2. Patient with documented HIV-1 infection
3. Subject has voluntarily signed and dated an informed consent form
4. Subject agrees not to take any medication during the study, including over the counter medicines or herbal preparations, without the approval of the trial physician.
5. Documented HIV-1 RNA >1,000 copies/mL
6. Subject naïve to ARV. (Patients who had received ARV ≤ 48 hours are allowed).
7. Subject has indication to receive an antiretroviral regimen.
8. Subjects can comply with protocol requirements.
9. Subject's general medical condition, in the investigator's opinion, does not interfere with assessments and completion of the trial.
10. If female, :

    1. use 2 different methods of birth control including, at least, one barrier method, and are acceptable to both the subject and investigator, and
    2. has a urine pregnancy test performed at the Screening Visit and on Baseline. Results of both tests must be negative.
    3. continue using 2 different methods of birth control including, at least, one barrier method for at least 30 days after the end of the treatment period

Exclusion Criteria:

* 1. Evidence of viral resistance against lopinavir/ritonavir, and/or FTC or 3TC, and/or other nucleoside analogues based on the genotype resistance test performed at screening, considering resistance according to the panel IAS - USA, version in December, 2009.

  2. The presence of any of the following major mutations: V32I; I47V / A; L76V; V82A/F/T/S or the presence of two or more minor mutations at positions:10,20,24,33,46,50,53,54,63,71,73,84,90 is considered resistance to lopinavir/ritonavir.

  3. The presence of mutation M184V/I and/or K65R is considered resistance to 3TC or FTC. At the discretion of the investigator and based on the resistance test, a treatment based on lopinavir / ritonavir, plus 3TC or FTC and other similar nucleoside / nucleotide active could not be constructed.

  4. Previously documented HIV-2 infection. 5. Use of disallowed concomitant therapy 6. Patient has a current (active) diagnosis of acute hepatitis due to any cause OR chronic Hepatitis C WITH aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >5 x upper limit of normal (ULN) AND/OR is likely to require treatment in the next year.

  7. Active Hepatitis B infection (regardless of stage of infection). 8. Any active clinically significant disease . 9. Subject has a currently active AIDS defining illness (Category C)30 days of screening. Subjects who are on stable maintenance therapy for an opportunistic infection may be enrolled.

  10. Life expectancy < 1 year according to the judgment of the investigator. 11. Screening laboratory analysis shows any of the following abnormal laboratory results:

  a. Hemoglobin < 8.0 g/dL b. Absolute neutrophil count < 750 cells/µL c. Platelet count < 50,000 mm3 d. Creatinine> 1.5 times the normal upper limit. 12. Subject enrolled in other clinical trials . 13. Use of any investigational agents within 30 days prior to screening. 14. Use of immunosuppressive drugs, cytokine inhibitors or other cytokines in the last year.

  15. Active substance use or abuse that the investigator determines may significantly interfere with study procedures 16. Any condition (including but not limited to alcohol and drug use) which in the opinion of the investigator, could compromise the subject's safety or adherence to the protocol.

  17. Subject is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
• Proportion of patients with HIV-1 RNA levels of less than 50 copies/mL in an intent-to-treat analysis at week 48 | 48 and 96 weeks

SECONDARY OUTCOMES:
• Proportion of patients with HIV-1 RNA levels of less than 400 copies/mL at week 24 and at week 48 | 48 weeks
  * Proportion of patients with HIV-1 RNA levels of less than 50 copies/mL at week 24.
  * Number and type of resistance mutations in case of virologic failure• CD4+ lymphocyte count and proportion evolution between baseline and week 24 and 48.
  * Comparison of lipid profiles after 48 weeks
  * Changes in quality of life, assessed by a validated questionnaire
  * Treatment survival and interruptions.
  * Frequency, type and severity of adverse events.
  * Frequency of opportunistic infections (OI) and disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Cahn, MD, PhD, Principal Investigator — FUNDACION HUESPED
Locations (1):
- Fundacion Huesped, Ciudad de Buenos Aires, Argentina

REFERENCES:
- [Derived] Cahn P, Andrade-Villanueva J, Arribas JR, Gatell JM, Lama JR, Norton M, Patterson P, Sierra Madero J, Sued O, Figueroa MI, Rolon MJ; GARDEL Study Group. Dual therapy with lopinavir and ritonavir plus lamivudine versus triple therapy with lopinavir and ritonavir plus two nucleoside reverse transcriptase inhibitors in antiretroviral-therapy-naive adults with HIV-1 infection: 48 week results of the randomised, open label, non-inferiority GARDEL trial. Lancet Infect Dis. 2014 Jul;14(7):572-80. doi: 10.1016/S1473-3099(14)70736-4. Epub 2014 Apr 27. PMID 24783988
- See also: Related Info — http://www.Huesped.org.ar/